CLINICAL TRIAL: NCT00164281
Title: A Randomized, Placebo-Controlled Study of Limited vs. Continuous Isoniazid Tuberculosis Preventive Therapy in HIV-infected Persons in Botswana
Brief Title: Study of Limited Versus Continuous Isoniazid Tuberculosis Preventive Therapy in HIV-infected Persons in Botswana
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Botswana Ministry of Health (Other Government); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-3441
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Tuberculosis; HIV Infections
Keywords: TB; Tuberculosis; INH; Isoniazid; Preventive therapy; HIV; AIDS; Botswana; LTBI; Latent TB Infection
MeSH Terms: conditions — Tuberculosis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Isoniazid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Continuous vs limited isoniazid (Experimental): The placebo arm will receive 6 months of open label isoniazid before beginning placebo (as a coded medication). The treatment (experimental arm) will receive 6 months of open label isoniazid before beginning coded medication (isoniazid).
  Interventions: Drug: Isoniazid

INTERVENTIONS:
Drug: Isoniazid — Daily 300 mg isoniazid supplemented with 25 mg pyridoxine for 6 months vs 36 months.
  Other Names: Isonicotinic Acid Hydrazide

SUMMARY:
This is a randomized, blinded, two-arm comparative trial of continued versus limited isoniazid (INH) tuberculosis (TB) preventive therapy in HIV-infected adults in Gaborone and Francistown, Botswana. Subjects will be accrued over two years and followed for a minimum of 36 months.

DETAILED DESCRIPTION:
Randomized, double blinded, two-arm comparative trial of continuous vs. limited isoniazid preventive therapy in HIV-infected adults in Gaborone and Francistown, Botswana. Subjects will be accrued over two years and followed for a minimum of 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected
2. Age >=18 years
3. Tuberculin skin test positive or negative
4. Laboratory:

   * Hemoglobin (Hgb) >6.5 gm/dl;
   * Neutrophil count >1,000 cells/mm3;
   * Platelets >75,000/mm3;
   * AST (SGOT) <122 U/L;
   * Creatinine <1.5 mg/dl;
   * Beta HCG = negative
5. Karnofsky performance status >=60
6. Signed informed consent

Exclusion Criteria:

1. History of TB in the last 3 years or current active TB
2. History of noncompliance to chronic therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2004-11; Primary Completion 2009-07 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Incident tuberculosis | During enrolment

SECONDARY OUTCOMES:
Death | During enrolment
Adverse events | During provision of study medication
  After enrolment, half of the participants will receive isoniazid for 6 months and the other half for 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Taraz Samandari, MD, PHD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Gaborone and Francistown Health Clinics, Gaborone and Francistown, Botswana

REFERENCES:
- [Background] Agizew T, Bachhuber MA, Nyirenda S, Makwaruzi VZ, Tedla Z, Tallaksen RJ, Parker JE, Mboya JJ, Samandari T. Association of chest radiographic abnormalities with tuberculosis disease in asymptomatic HIV-infected adults. Int J Tuberc Lung Dis. 2010 Mar;14(3):324-31. PMID 20132624
- [Background] Agizew TB, Arwady MA, Yoon JC, Nyirenda S, Mosimaneotsile B, Tedla Z, Motsamai O, Kilmarx PH, Wells CD, Samandari T. Tuberculosis in asymptomatic HIV-infected adults with abnormal chest radiographs screened for tuberculosis prevention. Int J Tuberc Lung Dis. 2010 Jan;14(1):45-51. PMID 20003694
- [Background] Mosimaneotsile B, Mathoma A, Chengeta B, Nyirenda S, Agizew TB, Tedla Z, Motsamai OI, Kilmarx PH, Wells CD, Samandari T. Isoniazid tuberculosis preventive therapy in HIV-infected adults accessing antiretroviral therapy: a Botswana Experience, 2004-2006. J Acquir Immune Defic Syndr. 2010 May 1;54(1):71-7. doi: 10.1097/QAI.0b013e3181c3cbf0. PMID 19934764
- [Background] Tedla Z, Nyirenda S, Peeler C, Agizew T, Sibanda T, Motsamai O, Vernon A, Wells CD, Samandari T. Isoniazid-associated hepatitis and antiretroviral drugs during tuberculosis prophylaxis in hiv-infected adults in Botswana. Am J Respir Crit Care Med. 2010 Jul 15;182(2):278-85. doi: 10.1164/rccm.200911-1783OC. Epub 2010 Apr 8. PMID 20378730
- [Result] Samandari T, Agizew TB, Nyirenda S, Tedla Z, Sibanda T, Shang N, Mosimaneotsile B, Motsamai OI, Bozeman L, Davis MK, Talbot EA, Moeti TL, Moffat HJ, Kilmarx PH, Castro KG, Wells CD. 6-month versus 36-month isoniazid preventive treatment for tuberculosis in adults with HIV infection in Botswana: a randomised, double-blind, placebo-controlled trial. Lancet. 2011 May 7;377(9777):1588-98. doi: 10.1016/S0140-6736(11)60204-3. Epub 2011 Apr 12. PMID 21492926
- [Result] Gust DA, Mosimaneotsile B, Mathebula U, Chingapane B, Gaul Z, Pals SL, Samandari T. Risk factors for non-adherence and loss to follow-up in a three-year clinical trial in Botswana. PLoS One. 2011 Apr 25;6(4):e18435. doi: 10.1371/journal.pone.0018435. PMID 21541021
- [Result] Chaisson LH, Kass NE, Chengeta B, Mathebula U, Samandari T. Repeated assessments of informed consent comprehension among HIV-infected participants of a three-year clinical trial in Botswana. PLoS One. 2011;6(10):e22696. doi: 10.1371/journal.pone.0022696. Epub 2011 Oct 27. PMID 22046230
- [Result] Sibanda T, Tedla Z, Nyirenda S, Agizew T, Marape M, Miranda AG, Reuter H, Johnson JL, Samandari T. Anti-tuberculosis treatment outcomes in HIV-infected adults exposed to isoniazid preventive therapy in Botswana. Int J Tuberc Lung Dis. 2013 Feb;17(2):178-85. doi: 10.5588/ijtld.12.0314. PMID 23317952
- [Result] Taylor AW, Mosimaneotsile B, Mathebula U, Mathoma A, Moathlodi R, Theebetsile I, Samandari T. Pregnancy outcomes in HIV-infected women receiving long-term isoniazid prophylaxis for tuberculosis and antiretroviral therapy. Infect Dis Obstet Gynecol. 2013;2013:195637. doi: 10.1155/2013/195637. Epub 2013 Mar 7. PMID 23533318
- [Derived] Tedla Z, Nguyen ML, Sibanda T, Nyirenda S, Agizew TB, Girde S, Rose CE, Samandari T. Isoniazid-associated hepatitis in adults infected with HIV receiving 36 months of isoniazid prophylaxis in Botswana. Chest. 2015 May;147(5):1376-1384. doi: 10.1378/chest.14-0215. PMID 25340318
- See also: Video webcast of preliminary results by Dr. T. Samandari on Feb 18, 2010 — http://www.retroconference.org/2010/data/files/webcast_2010.htm